CLINICAL TRIAL: NCT03392402
Title: Prospective Validation of the Molecular Classifier for the Fine Needle-based Assessment of Malignancy Risk in Thyroid Nodules
Brief Title: Molecular Classifier for the Fine Needle-based Assessment of Malignancy Risk in Thyroid Nodules
Acronym: ThyroPred-1
Status: Completed | Type: Observational
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 267398/4/NCBR/2015/1
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-07

CONDITIONS: Thyroid Nodule; Thyroid Neoplasm; Thyroid Cancer
Keywords: Thyroid nodule; Indeterminate thyroid nodule; Molecular biopsy; Gene expression classifier
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fine needle aspiration biopsy (FNAB) material and washout will be diluted in dedicated buffer and frozen in -80C. RNA and DNA will be isolated by commercial kits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the usefulness of molecular classifier to aid the diagnosis of malignancy in the material obtained by fine-needle aspiration biopsy (FNAB) of thyroid nodule. All participants will undergo FNAB with routine cytological assessment and molecular testing. Patients will undergo surgery or be followed-up, according to the clinical guidelines. The diagnostic power of combined molecular/clinical classifier will be compared to prediction based on clinical features only, by investigators blinded to the final diagnosis of surgical assessment.

DETAILED DESCRIPTION:
Currently, the diagnosis of malignancy of thyroid nodule is based on cytological assessment of fine-needle aspiration biopsy (FNAB) classified according to the Bethesda System for Reporting of Thyroid Cytopathology. This does not allow for the definitive diagnosis of cancer in significant proportion of tumors, so called indeterminate nodules (Bethesda class III, IV and V). These patients require surgery to establish a definitive diagnosis, leading to unnecessary operating procedures in at least 2/3 of subjects.

Molecular classifiers could significantly improve thyroid preoperative diagnostics, although they are not optimal and provide either high specificity to the detriment of low sensitivity or conversely, relatively low specificity with high sensitivity. The classifiers could be based on gene expression or mutations present in FNAB specimen.

In the present study the investigators plan to assess the improvement of classification power by molecular gene-expression-based multi-feature classifier when added to standard clinical parameters indicating the risk of malignancy (Bethesda class, tumor size, patient age and sex). Participants will undergo FNAB with prospective collection of material for molecular testing and simultaneous preoperative recording of all clinical parameters. The patients will be operated on or followed-up according to the clinical guidelines. The comparison of a predictive power of clinical criteria to the combined clinical-molecular classifier will be carried out by the group of investigators blinded to the results of final surgery.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of thyroid nodule
* considerable chance for surgical procedure following biopsy result
* patient's consent for collection of material during routine fine needle aspiration biopsy

Exclusion Criteria:

* age below 18 years
* the presence of contraindications that make surgical treatment impossible
* prior diagnosis of thyroid cancer
* antithrombotic treatment except of acetylsalicylic acid or low molecular weight heparin at a prophylactic dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (above 18 years old) diagnosed with a thyroid nodule, in whom the fine-needle aspiration biopsy is undertaken to establish the necessity of thyroid surgery
Sampling Method: Non-Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy in patients with indeterminate FNAB results who undergone surgery within 6 months from biopsy | until surgery or 6 months from biopsy
  The improvement in accuracy of classification will be compared between sole clinical criteria (Bethesda class, tumor size, age, and sex) and combined classifier built on both clinical parameters and gene expression data. The population of indeterminate nodules will be defined by expert analysis of cytological samples by pathologists blinded to the outcome of surgery. Diagnostic accuracy will defined as the percentage of patients who were correctly diagnosed as benign or malignant based on the data available preoperatively.

SECONDARY OUTCOMES:
Diagnostic accuracy in all patients recruited to the study, who were operated on or remained in follow-up for at least 24 months from biopsy. | until surgery or 24 months from biopsy
  The improvement in accuracy of classification will be compared between sole clinical criteria (Bethesda class, tumor size, age, and sex) and combined classifier built on both clinical parameters and gene expression data. All patients after surgery will be included. Tumors in patients not operated on will be considered benign after confirmation of stable tumor status at least with 24 months follow-up. Patients not operated on and with shorter follow-up will be excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Jarzab, MD, PhD, Study Chair — Maria Sklodowska-Curie National Research Institute of Oncology; Rafal Tarnawski, MD, PhD, Study Director — Maria Sklodowska-Curie National Research Institute of Oncology
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology, Gliwice, Poland

IPD SHARING:
Plan to Share IPD: Undecided